CLINICAL TRIAL: NCT00225719
Title: Regression of Coronary Atherosclerotic Lesions After rHDL Infusions in Acute Coronary Syndrome Patients as Assessed by Intravascular Ultrasound.
Brief Title: Effect of rHDL on Atherosclerosis - Safety and Efficacy: THE ERASE TRIAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Limited (Industry)
Responsible Party: Dr Russell Basser, CSL Limited
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSLCT-HDL-04-06
Record Dates: First submitted 2005-09-23; First posted 2005-09-26 (Estimated); Last update posted 2008-11-10 (Estimated); Status verified 2008-11

CONDITIONS: Acute Coronary Syndromes
MeSH Terms: conditions — Acute Coronary Syndrome

INTERVENTIONS:
Drug: rHDL

SUMMARY:
Currently available therapies to treat Acute Coronary Syndromes(ACS) have several limitations including; the relatively long treatment duration required before apparent significant benefit; the inability to achieve reversal of the atherosclerotic process; and poor patient compliance due to chronicity of therapy. This study will assess the effects of rHDL compared with placebo on indices of atherosclerosis progression and regression as assessed with intravascular ultrasound (IVUS) in patients after acute coronary syndromes (ACS).

ELIGIBILITY:
Inclusion Criteria:

* Male or female 30 - 75 years of age
* Recent acute coronary syndrome, defined as unstable angina, non-Q wave myocardial infarction, or ST elevation indicative of myocardial infarction, within the last 14 days

Exclusion Criteria:

* >50% stenosis by visual angiographic estimation in the left main artery
* Renal insufficiency
* Severe liver disease
* Congestive heart failure as defined by the NYHA classification as functional Class III or Class IV
* Previous or planned coronary artery bypass surgery

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2005-07

PRIMARY OUTCOMES:
Efficacy

SECONDARY OUTCOMES:
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Tardif, MD FRCP, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Tardif JC, Gregoire J, L'Allier PL, Ibrahim R, Lesperance J, Heinonen TM, Kouz S, Berry C, Basser R, Lavoie MA, Guertin MC, Rodes-Cabau J; Effect of rHDL on Atherosclerosis-Safety and Efficacy (ERASE) Investigators. Effects of reconstituted high-density lipoprotein infusions on coronary atherosclerosis: a randomized controlled trial. JAMA. 2007 Apr 18;297(15):1675-82. doi: 10.1001/jama.297.15.jpc70004. Epub 2007 Mar 26. PMID 17387133